CLINICAL TRIAL: NCT05537285
Title: Individualized Neuromodulation for Anhedonic Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Cornell University (Other); Stanford University (Other); Wellcome Leap Organization (Unknown)
Responsible Party: Principal Investigator, Zafiris Daskalakis, Professor of Psychiatry, Department Chair, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221649-2
Record Dates: First submitted 2022-08-04; First posted 2022-09-13 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: MDD; Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study will be evenly randomized into one of three treatment groups: Individualized Accelerated Intermittent Theta-Burst Stimulation (Ind-aiTBS), Standard aiTBS (Std-aiTBS). Treatments will last 1 week in all three arms.
Who Masked: Participant, Care Provider
Masking Description: Blinding will be achieved via a sham rTMS coil (Cool-B65 A/P) used with the device. This coil can deliver either active or sham stimulation in a manner that is randomized by the system itself and therefore blinded to the treater. The sham setting on this coil looks and sounds identical to the active setting but has a hidden aluminum plate blocking actual stimulation. The MagVenture TMS device holds a blinded key code that is kept by the individual that holds the blind. During the rTMS setup, the operator is instructed to flip the coil to correspond with the key code, but the operator is not able to discern the active versus sham stimulation. Additional measures will be taken to ensure that the treater remains blinded during treatment administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Individualized Accelerated Intermittent Theta Burst Stimulation (Ind-aiTBS) (Experimental): Patients will receive individualized unilateral accelerated theta-burst stimulation to the left dorsal lateral prefrontal cortex for 5 consecutive days, with a total of 10 hours a day. Treatment will be 10min with 50min of breaks in between the 10 sessions. The target for stimulation will be individualized using the participant's fMRI scans by finding the region of the DLPFC most anti-correlated with the subgenual anterior cingulate cortex (sgACC). This target will be determined using e-field modeling and theta-gamma coupling.
  Interventions: Device: Individualized Accelerated Intermittent Theta Burst Stimulation (Ind-aiTBS)
- Standard Accelerated Intermittent Theta Burst Stimulation (Std-aiTBS) (Active Comparator): Patients will receive unilateral accelerated theta-burst stimulation to the left dorsal lateral prefrontal cortex for 5 consecutive days, with a total of 10 hours a day. Treatment will be 10min with 50min of breaks in between the 10 sessions.
  Interventions: Device: Standard Accelerated Intermittent Theta Burst Stimulation (Std-aiTBS)
- Sham Accelerated Intermittent Theta Burst Stimulation (sham) (Sham Comparator): Patients will receive sham unilateral accelerated theta-burst stimulation to the left dorsal lateral prefrontal cortex for 5 consecutive days, with a total of 10 hours a day. Treatment will be 10min with 50min of breaks in between the 10 sessions.
  Interventions: Device: Sham Accelerated Intermittent Theta Burst Stimulation (Sham)

INTERVENTIONS:
Device: Individualized Accelerated Intermittent Theta Burst Stimulation (Ind-aiTBS) — active side magnetic coil stimulation applied to individualized target in the left dorsal lateral prefrontal cortex.
  Other Names: MagStim Cool B65- A/P
  Arms: Individualized Accelerated Intermittent Theta Burst Stimulation (Ind-aiTBS)
Device: Standard Accelerated Intermittent Theta Burst Stimulation (Std-aiTBS) — active side magnetic coil stimulation applied to standardized target in the left dorsal lateral prefrontal cortex.
  Other Names: MagStim Cool B65- A/P
  Arms: Standard Accelerated Intermittent Theta Burst Stimulation (Std-aiTBS)
Device: Sham Accelerated Intermittent Theta Burst Stimulation (Sham) — sham side magnetic coil stimulation applied to the left dorsal lateral prefrontal cortex.
  Other Names: MagStim Cool B65- A/P
  Arms: Sham Accelerated Intermittent Theta Burst Stimulation (sham)

SUMMARY:
This program of research constitutes a three-arm, randomized, placebo-controlled trial testing noninvasive brain stimulation for the treatment of anhedonic depression. This trial is part of a larger, three-site study that will be conducted at UCSD, Stanford University, and Cornell University, with the overarching goals to compare competing interventions tested at each site and to combine data that will allow for the creation of an end-to-end model of anhedonic depression. By doing this, the investigators hope to gain insight and lead to the development of brain-behavior biomarkers to identify who is best suited for the different treatment options tested at each site. An additional exploratory objective is phenotyping anhedonic depression from the acquired measures.

Anhedonic patients recruited at UCSD will be randomized to one of three treatment arms to receive different forms of accelerated intermittent theta burst stimulation (aiTBS),a novel form of repetitive transcranial magnetic stimulation (rTMS) that is an FDA approved treatment for depression. These arms include: individualized accelerated iTBS (Ind-aiTBS),based on both the frequency of brain responses and electric-field (e-field) modeling of brain bioconductivity; standard accelerated iTBS (Std-aiTBS); and accelerated sham iTBS(sham). Treatment will be delivered on an accelerated schedule, over one week. Additional study sessions will occur both before and after treatment to assess for clinical, neurophysiological, and cognitive measures that will allow for both individualization of treatment and detailed assessment of the effects of the different treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, between the ages of 18 and 80 at the time of screening.
* Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questionnaires / follow instructions during fMRI assessments and aiTBS interventions. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
* Currently diagnosed with Major Depressive Disorder (MDD) or Bipolar Disorder type II and meets criteria for a Major Depressive Episode, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
* Medical records confirming a history of moderate to severe treatment-resistance as defined an Antidepressant Treatment History Form (ATHF) score for that antidepressant trial of > 3 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF score of 1 or 2 on those 2 separate antidepressants) OR have a combination of one failed trial and one not tolerated trial, per the definitions above.
* MADRS score of ≥20 at screening (Visit 1).
* Access to ongoing psychiatric care before and after completion of the study.
* Access to open label neuromodulation treatment after study completion.
* Must be on a stable antidepressant therapeutic regimen for 6 weeks prior to study enrollment and agree to continue this regimen throughout the study period.
* In good general health, as evidenced by medical history.
* For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
* Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

* Pregnancy
* History of or current psychotic disorder or depression with psychotic features
* Severe borderline personality disorder.
* Diagnosis of Intellectual Disability or Autism Spectrum Disorder
* Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
* Urine screening test positive for illicit substances
* Clinically significant suicidal ideation with plan
* Any history of ECT (greater than 8 sessions) without a clinical meaningful response.
* Recent (during the current depressive episode) or concurrent use of rapid acting antidepressant agent (i.e., ketamine or a course of ECT) in the last 30 days
* History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
* Untreated or insufficiently treated endocrine disorder.
* Contraindication to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
* Contraindication to MRI (ferromagnetic metal in their body)
* Treatment with an investigational drug or other intervention within the study period
* Unstable symptoms between screening and baseline as defined by a ≥ 30% change in MADRS score.
* Require a benzodiazepine with a dose > lorazepam 2 mg/day or equivalent or any anticonvulsant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS Scores | 8 weeks
  To evaluate the effects of individualized accelerated iTBS (using BOTH the frequency and e-field individualization; Ind-aiTBS) compared to standard accelerated iTBS (Std-aiTBS) and sham accelerated iTBS (sham) on depression severity measured with the Montgomery- Asbery Depression Rating Scale (MADRS).
Change in DARS Scores | 8 weeks
  To evaluate the effects of individualized accelerated iTBS (using BOTH the frequency and e-field individualization; Ind-aiTBS) compared to standard accelerated iTBS (Std-aiTBS) and sham accelerated iTBS (sham) on anhedonia as measured with the Dimensional Anhedonia Rating Scale (DARS).

SECONDARY OUTCOMES:
Assessment of Neuroplasticity | 8 weeks
  Analysis of transcranial magnetic stimulation concurrent with electroencephalogram (TMS-EEG) to extract activation of the left dorsolateral prefrontal cortex (DLPFC). Changes in activation between pre- and post-neurophysiology measures will be compared between the three treatment arms to determine the effects of Ind-aiTBS on neuroplasticity as compared to Std-aiTBS and sham.

OTHER OUTCOMES:
Predictive TMS-EEG Biomarker | 8 weeks
  Determine if baseline TMS-EEG predicts changes in anhedonia symptoms, as measured through correlation with changes in the MADRS and DARS from pre- to post-treatment.
Predictive fMRI Biomarker | 8 weeks
  Determine if baseline fMRI predicts changes in anhedonia symptoms, as measured through correlation with changes in the MADRS and DARS from pre- to post-treatment.
Cross-Sectional TMS-EEG Biomarker | 8 weeks
  Test for cross-sectional differences in TMS-EEG as a function of anhedonia symptoms measured by the MADRS and DARS at pre-treatment.
Cross-Sectional fMRI Biomarker | 8 weeks
  Test for cross-sectional differences in fMRI as a function of anhedonia symptoms measured by the MADRS and DARS at pre-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Interventional Psychiatry, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No